CLINICAL TRIAL: NCT06770257
Title: A Randomized Phase ll Study Evaluating the Efficacy and Safety of Combination Therapy of Daunorubicin, Cytarabine Liposomes and Venetoclax Versus Combination Therapy of Azacitidine and Venetoclax in Newly Diagnosed AML Patients Not Eligible for Intensive Chemotherapy
Brief Title: Daunorubicin, Cytarabine Liposomes Plus Venetoclax vs Azacitidine Plus Venetoclax in AML Patients Unfit for Intensive Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The project was terminated as the genetic office did not approve it.
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024082
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ArmA（daunorubicin, cytarabine liposomes plus 14d-venetolcax） (Experimental): Patients receive daunorubicin, cytarabine liposomes through intravenous injection(IV) on days 1、3、5, and venetoclax orally（PO） daily on days 1-14. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: daunorubicin, cytarabine liposomes; Drug: Venetoclax
- ArmB（daunorubicin, cytarabine liposomes plus 28d-venetolcax） (Experimental): Patients receive daunorubicin, cytarabine liposomes IV on days 1、3、5, and venetoclax PO daily on days 1-28. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: daunorubicin, cytarabine liposomes; Drug: Venetoclax
- ArmC（azacitidine plus 28d-venetoclax） (Active Comparator): Patients receive azacitidine subcutaneously (SC) on days 1-7, and venetoclax PO daily on days 1-28. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: daunorubicin, cytarabine liposomes — First induction: 100 units/m^2 by 90-minute IV infusion on Days 1, 3, 5. Second induction: 100 units/m^2 by 90-minute IV infusion on Days 1 and 3. Consolidation therapy: 65 units/m^2 by 90-minute IV infusion on Days 1 and 3.
  Arms: ArmA（daunorubicin, cytarabine liposomes plus 14d-venetolcax）; ArmB（daunorubicin, cytarabine liposomes plus 28d-venetolcax）
Drug: Azacitidine — Given SC on days 1-7
  Arms: ArmC（azacitidine plus 28d-venetoclax）
Drug: Venetoclax — Given PO on days 1-14 or 1-21 or 1-28

SUMMARY:
Daunorubicin, Cytarabine Liposomes(CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd.) is a dual-drug liposomal encapsulation of cytarabine and daunorubicin at a fixed 5:1 synergistic molar ratio.

This is a phase 2, randomized, controlled study in patients who are >= 18 or more years old and have not been treated before. Participants who take part in this study should not be suitable for intensive induction therapy.

In this study, patients will be randomized by 1:1:1 to receive Daunorubicin, Cytarabine Liposomes + Venetoclax(14d) or Daunorubicin, Cytarabine Liposomes + Venetoclax(21d) or Venetoclax + Azacitidine.

Participants will continue to have study visits and receive treatment for as long as they are having a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have confirmation of Acute Myeloid Leukemia (AML) by 2022 World Health Organization (WHO) criteria, previously untreated.
2. Participant must be >= 18 years of age.
3. Participant must have a projected life expectancy of at least 12 weeks.
4. Participant must be considered ineligible for intensive induction therapy defined by the following:

   a. >= 75 years of age; b. >= 18 to 74 years of age with at least one of the following comorbidities: i. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3; ii. Cardiac history of Congestive Heart Failure (CHF) requiring treatment or Ejection Fraction <= 50% or chronic stable angina; iii. Diffusing capacity of the Lung for Carbon Monoxide (DLCO) <= 65% or Forced Expiratory Volume in 1 second (FEV1) <= 65%; iv. Creatinine clearance >= 30 mL/min to < 45 ml/min; v. Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × Upper Limit of Normal (ULN); vi. Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy.
5. Participant must have an ECOG Performance status:

0 to 2 for Participants >= 75 years of age or 0 to 3 for Participants >= 18 to 74 years of age. 6.Laboratory values meet the following criteria:

1. Serum alanine aminotransferase or aspartate aminotransferase≤3 × ULN, ≤5 × ULN for patients with liver involvement.
2. For participants of ≥ 75 years old: Serum total bilirubin≤1.5 × ULN, ≤3 × ULN for patients with liver involvement
3. For participants of 18 to 74 years old: Serum total bilirubin≤ 3× ULN
4. Adequate renal function as demonstrated by a creatinine >= 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.

   7.Male participants who are sexually active, must agree, from Study Day 1 through at least 6 months after the last dose of study drug, to practice the protocol specified contraception and agree to refrain from sperm donation during this period.

   8.Female participants of childbearing potential must practice the protocol specified contraception from Study Day 1 through at least 6 months after the last dose of study drug. Female participants must agree to refrain from preganancy, breastfeeding or egg donation during this period. Female participants of childbearing potential must have negative results for pregnancy test performed: At Screening with a serum sample obtained within 7 days prior to the first study drug administration.

   9.Participant must able to understand the study and voluntarily sign informed consent.

   -

   Exclusion Criteria:
   1. White blood cell count>25 × 10 ^ 9/L (treatment with hydroxyurea or leukocyte isolation is allowed);
   2. Acute promyelocytic leukemia (APL);
   3. Previously received treatment with vinaclor or demethylating drugs or other chemotherapy drugs for AML or MDS (excluding the use of hydroxyurea before study administration)
   4. AML participants with good cytogenetic characteristics, including T (8; 21)/RUNX1:: RUNX1T1 or inv16/CBFB:: MYH11；
   5. AML secondary to MPN (including myelofibrosis, polycythemia vera, primary thrombocytosis, CML) and accompanied by BCR: AML participants of ABL1;
   6. AML participants with known central nervous system involvement;
   7. Within 6 months prior to the first administration, there is active cardiovascular disease, including but not limited to the following conditions: myocardial infarction, unstable angina, uncontrolled arrhythmia, and grade III/IV heart failure (New York Heart Association standard, NYHA); Hypertension that is still poorly controlled after antihypertensive treatment (with three consecutive measurements of systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 90mmHg during the screening period).
   8. hepatitis B B surface antigen (HBsAg) positive/hepatitis B B core antibody (HBcAb) positive, HBV DNA higher than the measurable lower limit or 1000 copies/mL (500IU/mL) (whichever is lower), HCV antibody positive and HCV RNA higher than the measurable lower limit or 1000 copies/mL (whichever is lower);
   9. History of immunodeficiency, including positive HIV antibody test;
   10. Have used other clinical trial drugs for treatment within one month before receiving treatment;
   11. Participants who received potent or moderate cytochrome P450 3A (CYP3A) inducers/inhibitors or P-glycoprotein (P-gp) inhibitors within 7 days prior to commencing study treatment;
   12. Participants have consumed grapefruit, grapefruit products, Seville oranges (including jam containing Seville oranges), or starfruit within 3 days prior to the first administration of the study drug.
   13. Have a history of allergic reactions to the ingredients of the research drug (and its excipients) and/or other similar products;
   14. Wilson's disease history or other history of copper metabolism abnormalities;
   15. Participants with cumulative exposure to anthracycline drugs exceeding 339 mg/m2 of daunorubicin (or equivalent drug dose level);
   16. Pregnancy or lactation period;
   17. Participants who are unable to take oral medication, have malabsorption syndrome, or suffer from other diseases that hinder enteral administration;
   18. Uncontrolled active infections (viruses, bacteria, or fungi) (the infection must be controllable for at least 3 consecutive days with normal body temperature and stable hemodynamics in co infected participants using antibiotics)
   19. History of other malignant tumors within the past 3 years or concurrent active malignant tumors, excluding: 1) cervical carcinoma in situ or breast carcinoma in situ that has received adequate treatment; 2) basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; 3) localized malignant tumors that have been surgically removed (or treated in other ways) for the purpose of cure;
   20. Suffer from any serious and/or uncontrollable disease that may affect the participants' participation in this study as determined by the investigator (including but not limited to chronic respiratory disease requiring continuous oxygen inhalation, diabetes not effectively controlled, kidney disease requiring dialysis, serious liver disease, life-threatening autoimmune disease and hemorrhagic disease, drug abuse, nervous system disease, etc.);
   21. There are other situations deemed unsuitable by the researchers to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate(CR) | Up to 8 months
  Proportion of patients with complete remission during the treatment period.

SECONDARY OUTCOMES:
Composite complete remission rate(cCR) | Up to 8 months
  Proportion of CR and complete remission with incomplete count recovery(CRi)
Proportion of pateints who achieve Measurable residual disease（MRD） negativity | Up to 8 months
  The percentage of patients who are MRD negative
Event-free survival (EFS) | Up to 2 years
  EFS is defined as the time from study randomization to the date of induction treatment failure, disease relapse or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival will be measured from the date of randomization to death from any cause.